CLINICAL TRIAL: NCT02032511
Title: Comparison of RAM Cannula NCPAP Versus Infant Flow NCPAP
Brief Title: Comparison of RAM Cannula Nasal Continuous Positive Airway Pressure Versus Infant Flow Nasal Continuous Positive Airway Pressure (NCPAP)
Status: Terminated | Type: Observational
Why Stopped: No appreciable difference noted between methods of delivery
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michelle Pape, RRT, University of Michigan
Other Study IDs: HUM00073557
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Acute Respiratory Deficiency; Prematurity; Assisted Ventilation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RAM Cannula Nasal Continuous Positive Airway Pressure
- Infant Flow Nasal Continuous Positive Airway Pressure (NCPAP)

SUMMARY:
This study is designed to compare the effectiveness and ease of use of two commonly used NCPAP interfaces: the RAM NC and the Infant Flow prongs and nasal mask.

ELIGIBILITY:
Inclusion Criteria:

* less than or equal to 7 kg
* order for nasal continuous positive pressure

Exclusion Criteria:

* patients greater than 7kg
* patients that do not have informed consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants less than or equal to 7kg with an order for nasal continuous positive pressure
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of patients who achieve unassisted breathing | One year